CLINICAL TRIAL: NCT01448434
Title: A Randomized, Double Blind, Multicentric, Placebo Controlled, Phase -II Study Assessing the Safety and Efficacy of Intraarticular Ex-vivo Cultured Adult Allogeneic Mesenchymal Stem Cells in Patients With Osteoarthritis of Knee
Brief Title: Allogeneic Mesenchymal Stem Cells for Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stempeutics Research Pvt Ltd (Industry)
Collaborators: Stempeutics Research Malaysia SDN BHD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SRM/OA/10-11/001
Record Dates: First submitted 2011-09-20; First posted 2011-10-07 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Osteoarthritis of Knee Joint
Keywords: Osteoarthritis; Knee; Stem cell; MSC
MeSH Terms: conditions — Osteoarthritis | interventions — Plasmalyte A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ex- vivo cultured adult allogeneic MSCs (Experimental): Single intraarticular dose of allogeneic MSCs
  Interventions: Biological: Ex- vivo cultured adult allogeneic MSCs
- Plasmalyte-A (Placebo Comparator): Single intraarticular dose of 2ml Plasmalyte
  Interventions: Biological: Plasmalyte-A

INTERVENTIONS:
Biological: Ex- vivo cultured adult allogeneic MSCs — Single intraarticular dose of allogeneic MSCs suspended in 2ml Plasmalyte followed by 2ml of Hyaluronan
  Arms: Ex- vivo cultured adult allogeneic MSCs
Biological: Plasmalyte-A — Single intraarticular dose of 2ml Plasmalyte followed by 2ml Hyaluronan
  Arms: Plasmalyte-A

SUMMARY:
This study is designed to know the safety and efficacy of 2 different doses of mesenchymal stem cells in patients suffering from osteoarthritis of knee joint.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females in the age 20 - 70 years (both inclusive)
2. Radiographic evidence of grade 2 to 3 osteoarthritis based on the Kellgren and Lawrence radiographic entry criteria.
3. History of primary idiopathic osteoarthritis of the knee characterized by pain which requires intake of analgesics.
4. Self-reported difficulty in at least one of the following activities attributed to knee pain: lifting and carrying groceries, walking 400 metres, getting in and out of a chair, or going up and down stairs.
5. Patients who have been on stable medication for the past three months.
6. Patients who have not received intra articular steroids or hyaluronan within the last three months.
7. Female patients of childbearing age must be willing to use accepted methods of contraception during the course of the study
8. Ability to provide written informed consent.

Exclusion Criteria:

1. Prior or ongoing medical conditions (e.g., concomitant illness, psychiatric condition, alcoholism, drug abuse), medical history, physical findings, ECG findings, or laboratory abnormality that, in the investigator's opinion, could adversely affect the safety of the subject, makes it unlikely that the course of treatment or follow-up would be completed, or could impair the assessment of study results.
2. History of surgery, including arthroscopy, or major trauma to the study joint in the previous 12 months
3. Signs of active study joint inflammation including redness, warmth, and/or, if qualifying with osteoarthritis of the knee, a large, bulging effusion of the study knee joint with the loss of normal contour of the joint at the screening visit or at the baseline examination
4. Infections in or around the knee.
5. Patients awaiting a replacement knee or hip joint
6. Patients with other conditions that cause pain
7. Significantly incapacitated or disabled and would be categorized as ACR Functional Class IV (largely or wholly incapacitated), or unable to walk without assistive devices
8. Patients with other known rheumatic or inflammatory disease such as rheumatoid arthritis
9. Other pathologic lesions on x-rays of knee
10. Positive hepatitis B surface antigen, hepatitis C antibody test, Anti human immunodeficiency virus (HIV) antibody test, or VDRL
11. History of Bleeding disorders
12. Known hypersensitivity to Hyaluronan products or animal sera
13. For women of child-bearing potential: positive pregnancy test or lactating

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Number and percentage of patients with adverse events as a measure of safety and tolerability | 1 year
  * Safety evaluation will include assessment of physical examination, periodic monitoring of vital signs (heart rate, respiratory rate, blood pressure and temperature), clinical laboratory investigations (including haematology, serum chemistry, LFT, urine-analysis) and 12-lead ECG recording.
  * Tolerability: Adverse events monitored using information volunteered by the patients and as observed by the PI will be summarized descriptively by total number of AE(s) and compared between the study arms.

SECONDARY OUTCOMES:
Change from baseline in the WOMAC OA (Western Ontario and McMaster Universities Osteoarthritis) Index -pain subscale score | 1 Year
Change from baseline in WOMAC OA stiffness index | 1 Year
Change from baseline in WOMAC OA composite index | 1 Year
Change from baseline in ICOAP (Intermittent and Constant Osteoarthritis Pain) | 1 Year
Change from baseline in radiographic (X-ray) findings of knee | 1 Year
Change from baseline in the WORMS score of knee using MRI | 1 Year
Change from baseline in arthritis pain scores on the visual analogue scale | 1 Year
Reduction in the intake of analgesic tablets from baseline | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Muhammad Ali Noor Muhd Abdul Ghani, FRCS, Principal Investigator — KPJ Ampang Puteri Specialist Hospital; Dr. Ahmad Hisham Abd. Rashid, MD., MS, Principal Investigator — Clinical Research Centre Hospital Serdang; Dr. Suntharalingam Subramaniam, FRCS, Principal Investigator — Pantai Cheras Medical Centre; Dato' Dr. Ramli Baba, MS, Principal Investigator — Selayang Hospital
Locations (4):
- Malaysia (4):
  - Pantai Cheras Medical Centre, Kuala Lumpur, Kuala Lumpur
  - Serdang Hospital, Kuala Lumpur, Selangor
  - KPJ Ampang Puteri Specialist Hospital, Kuala Lumpur, Selangor
  - Selayang Hospital, Kuala Lumpur, Selangor